CLINICAL TRIAL: NCT03434015
Title: Post-approval Study of Percutaneous Left Atrial Appendage Closure
Brief Title: Post-approval Study of Percutaneous Left Atrial Appendage Closure ( FLAAC-2 )
Acronym: FLAAC-2
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 3528-NI
Record Dates: First submitted 2018-01-25; First posted 2018-02-15 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Left atrial septal closure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Left atrial appendage closure: All patient referred to a department of interventional cardiology for percutaneous left atrial appendage closure may be included.
  All centers practicing this procedure in France will participate to the present study, whatever the technique used. The patients included in the protocol will be followed as part of the care by centers that will have carried out the procedure.

SUMMARY:
Patients with atrial fibrillation are at significant risk of thrombus formation in the left atrial appendage, which can lead to a stroke or systemic embolism. This risk justifies first-line prescribing of long-term oral anticoagulant therapy in these patients. Percutaneous left atrial appendage closure, is a new interventional cardiology technique for patients at high risk of stroke related to atrial fibrillation in whom long term anticoagulation therapy cannot be conducted. This procedure involves implantation of an occlusion device into the left atrial appendage to close it and prevent migration of thrombotic material that can cause distant embolism. Closure of the left atrial appendage avoids long term prescription of anticoagulants while protecting patients against the risk of systemic embolism and stroke. In 2016, two devices developed for transcutaneous closure of the left atrial appendage (WATCHMAN, Boston Scientific, AMPLATZER CARDIAC PLUG, S. Jude Medical and its evolution AMPLATZER AMULET) were included in the list of products reimbursable in France. The French national authorities have requested the realization of a register whose objectives will be to evaluate:

* The efficiency and safety of implanting devices in France
* The type and duration of antithrombotic treatment prescribed after left atrial appendage closure

ELIGIBILITY:
Inclusion Criteria:

Any patient for whom an indication has been made for implantation of a device for the closure of the left atrial appendage without restriction of indication and regardless of the outcome of the procedure (implantation success or not).ot).

Exclusion Criteria:

* Refusal of the patient to participate in this study and therefore the use of his data
* Minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All French centers practicing percutaneous closure of the left atrial appendage will participate in the present study, whatever the technique used. The patients included in the protocol will be followed as part of the care by the centers that will have carried out the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Frequency of events at one year | 1 year
  The primary efficacy endpoint is the frequency of a combined endpoint including ischemic strokes, systemic embolism, unexplained deaths, and cardiovascular death one year after left atrial appendage closure. This frequency will be expressed as the percentage of patients who presented at least one of these events. Only the first event occurring in each patient concerned will be taken into account, in the case where the same patient would present several events.

SECONDARY OUTCOMES:
Efficacy at the end of the procedure | One hour after the end of the procedure
  At the end of the procedure, the efficiency of the procedure will be described by the percentage of success of the procedure. The successful procedure is defined by a successful implantation of the device in the left atrial appendage without presaging its occlusive character.
Percentage of occlusion of the left atrial appendage objectified by transesophageal echography at 3 months of follow up | 3 months of follow up
  Percentage of patients in whom the left atrial appendage is effectively closed,
Percentage of residual leakage revealed by transesophageal echocardiography at 3 months of follow up | 3 months of follow up
  Percentage of patients with residual leakage
Percentage of ischemic stroke at 1 year of follow up | 1 year of follow up
  Percentage of patients with at least one ischemic stroke between the procedure and the 1-year visit
Percentage of transient ischemic attack (TIA) at 1 year of follow up | 1 year of follow up
  Percentage of patients presenting at least one TIA between the procedure and the 1-year visit
Percentage of systemic embolism at 1 year of follow up | 1 year of follow up
  Percentage of patients with at least one systemic embolism between procedure and follow-up at 1 year
Percentage of cardiovascular or unexplained death at 1 year of follow up | 1 year of follow up
  Percentage of patients who had a cardiovascular or unexplained death between the procedure and the 1-year follow-up
Mortality at 1 year of follow up | 1 year of follow up
  Percentage of deaths between procedure and follow-up at 1 year
Frequency of cerebral or systemic ischemic events at 1 year of follow up | 1 year of follow up
  Comparison of the frequency of cerebral or systemic ischemic events to the predicted theoretical value according to the CHA2DS2-VASc score of the population included
Rate of complications related or potentially related to the device or the implantation procedure after 7 days of follow up | 7 days of follow up or discharge (if later then D7)
  Rate of complications related or potentially related to the device or the implantation procedure
Percentage of pericardial effusion after 7 days of follow up | 7 days of follow up or discharge (if later then D7)
  Percentage of patients who presented a pericardial effusion objectified by trans-thoracic ultrasound between the procedure and the discharge from hospital
Percentage of migration of the device after 7 days of follow up | 7 days of follow up or discharge (if later then D7)
  Percentage of patients who presented a migration of the device, objectified by the trans-thoracic ultrasound between the procedure and discharge
Percentage of device thrombosis at 3 months of follow up | 3 months of follow up
  Percentage of patients who presented thrombosis on the device, objectified by transesophageal echography and / or CT scan
Percentage of device migration at 3 months of follow up | 3 months of follow up
  Percentage of patients who had a migration of the device, objectified by transesophageal echography and / or CT scan
Rate of complications related or potentially related to the device or procedure after 1 year of follow up | 1 year of follow up
  Percentage of patients who had at least one device or procedure complication, such as tamponade requiring surgical drainage, device migration, residual leakage between procedure and 1 year follow-up
Device thrombosis or device migrations by trans-thoracic ultrasound after 1 year of follow up | 1 year of follow up
  Percentage of device thrombosis or device migrations by trans-thoracic ultrasound
Clinical evolution of the patient at 1 year | 1 year of follow up
  The percentage of life threatening, disabling or major hemorrhagic complications that occurred between the procedure and the 1-year follow-up will be recorded.
Criteria for Evaluating Associated Antithrombotic Treatments | 1 year of follow up
  The antithrombotic treatments will be collected at patient's exit, and at 3, 6 and 12 months after implantation.
  The type and duration of anti-thrombotic treatments will be documented using the combined criteria:
  * Percentage of patients on injectable or oral anticoagulants and antiplatelet agents at different follow-up times
  * Percentage of patients on injectable or oral anticoagulants at different follow-up times
  * The percentage of patients on platelet antiaggregants in single or dual therapy at different follow-up times
  * The average duration of anticoagulant and antiplatelet treatments
Description of the population and centers | At inclusion
  Demographic and clinical characteristics of the patients will be collected and described, such as: age, sex, medical and surgical history, cardiovascular pharmacological treatments, comorbidities, indication of left atrial closure, HAS-BLED and CHA2DS2-VASc scores, anatomical features of the left atrial appendage at inclusion.
  The type of health facility and the profile of the investigators will be evaluated according to:
  * The place of exercise of the investigators: percentage of physicians practicing in public centers, percentage of physicians practicing in hospital, percentage of physicians practicing in the private sector, percentage of physicians practicing in two sectors
  * The average number of implantations of each device made by the investigators since their first use of each system
Evaluation of implantation indications | At inclusion
  The cause of left atrial appendage closure will also be evaluated by comparing the indications of implantation of the device with the indications retained by the CNEDIMTS, taking into account the following combined criteria:
  * CHA2DS2-VASc Score
  * Strict contraindication to anticoagulant therapy
  * Nonvalvular FA

CONTACTS AND LOCATIONS:
Overall Officials: Nicole NACCACHE, Study Chair — French Society of Cardio
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Menke J, Luthje L, Kastrup A, Larsen J. Thromboembolism in atrial fibrillation. Am J Cardiol. 2010 Feb 15;105(4):502-10. doi: 10.1016/j.amjcard.2009.10.018. PMID 20152245
- [Background] Feinberg WM, Blackshear JL, Laupacis A, Kronmal R, Hart RG. Prevalence, age distribution, and gender of patients with atrial fibrillation. Analysis and implications. Arch Intern Med. 1995 Mar 13;155(5):469-73. PMID 7864703
- [Background] Heeringa J, van der Kuip DA, Hofman A, Kors JA, van Herpen G, Stricker BH, Stijnen T, Lip GY, Witteman JC. Prevalence, incidence and lifetime risk of atrial fibrillation: the Rotterdam study. Eur Heart J. 2006 Apr;27(8):949-53. doi: 10.1093/eurheartj/ehi825. Epub 2006 Mar 9. PMID 16527828
- [Background] Knecht S, Wilton SB, Haissaguerre M. The 2010 update of the ESC guidelines for the management of atrial fibrillation. Circ J. 2010 Nov;74(12):2534-7. doi: 10.1253/circj.cj-10-1030. Epub 2010 Nov 2. No abstract available. PMID 21060205
- [Background] Blackshear JL, Odell JA. Appendage obliteration to reduce stroke in cardiac surgical patients with atrial fibrillation. Ann Thorac Surg. 1996 Feb;61(2):755-9. doi: 10.1016/0003-4975(95)00887-X. PMID 8572814
- [Background] Lam YY, Yip GW, Yu CM, Chan WW, Cheng BC, Yan BP, Clugston R, Yong G, Gattorna T, Paul V. Left atrial appendage closure with AMPLATZER cardiac plug for stroke prevention in atrial fibrillation: initial Asia-Pacific experience. Catheter Cardiovasc Interv. 2012 Apr 1;79(5):794-800. doi: 10.1002/ccd.23136. Epub 2011 Nov 30. PMID 21542102
- [Background] Dawson AG, Asopa S, Dunning J. Should patients undergoing cardiac surgery with atrial fibrillation have left atrial appendage exclusion? Interact Cardiovasc Thorac Surg. 2010 Feb;10(2):306-11. doi: 10.1510/icvts.2009.227991. Epub 2009 Nov 26. PMID 19942634
- [Background] Sievert H, Lesh MD, Trepels T, Omran H, Bartorelli A, Della Bella P, Nakai T, Reisman M, DiMario C, Block P, Kramer P, Fleschenberg D, Krumsdorf U, Scherer D. Percutaneous left atrial appendage transcatheter occlusion to prevent stroke in high-risk patients with atrial fibrillation: early clinical experience. Circulation. 2002 Apr 23;105(16):1887-9. doi: 10.1161/01.cir.0000015698.54752.6d. PMID 11997272
- [Background] Klug D, Commeau P, Defaye P, Thambo JB, Gras D, Aubry P, Pasquie JL, Guerin P, Teiger E, Koning R, Piot O; Heart Rhythm, Pacing Group, the Atheroma, Interventional Cardiology Group of the French Society of Cardiology. Percutaneous occlusion of the left atrial appendage: An expert consensus statement. Arch Cardiovasc Dis. 2015 Aug-Sep;108(8-9):460-7. doi: 10.1016/j.acvd.2015.02.001. PMID 26645055
- [Background] Park JW, Bethencourt A, Sievert H, Santoro G, Meier B, Walsh K, Lopez-Minguez JR, Meerkin D, Valdes M, Ormerod O, Leithauser B. Left atrial appendage closure with Amplatzer cardiac plug in atrial fibrillation: initial European experience. Catheter Cardiovasc Interv. 2011 Apr 1;77(5):700-6. doi: 10.1002/ccd.22764. Epub 2011 Mar 8. PMID 20824765
- [Background] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Background] Belgaid DR, Khan Z, Zaidi M, Hobbs A. Prospective randomized evaluation of the watchman left atrial appendage closure device in patients with atrial fibrillation versus long-term warfarin therapy: The PREVAIL trial. Int J Cardiol. 2016 Sep 15;219:177-9. doi: 10.1016/j.ijcard.2016.06.041. Epub 2016 Jun 15. PMID 27343417
- [Background] Boersma LV, Schmidt B, Betts TR, Sievert H, Tamburino C, Teiger E, Pokushalov E, Kische S, Schmitz T, Stein KM, Bergmann MW; EWOLUTION investigators. Implant success and safety of left atrial appendage closure with the WATCHMAN device: peri-procedural outcomes from the EWOLUTION registry. Eur Heart J. 2016 Aug;37(31):2465-74. doi: 10.1093/eurheartj/ehv730. Epub 2016 Jan 27. PMID 26822918
- [Background] Holmes DR, Reddy VY, Turi ZG, Doshi SK, Sievert H, Buchbinder M, Mullin CM, Sick P; PROTECT AF Investigators. Percutaneous closure of the left atrial appendage versus warfarin therapy for prevention of stroke in patients with atrial fibrillation: a randomised non-inferiority trial. Lancet. 2009 Aug 15;374(9689):534-42. doi: 10.1016/S0140-6736(09)61343-X. PMID 19683639
- [Background] Reddy VY, Mobius-Winkler S, Miller MA, Neuzil P, Schuler G, Wiebe J, Sick P, Sievert H. Left atrial appendage closure with the Watchman device in patients with a contraindication for oral anticoagulation: the ASAP study (ASA Plavix Feasibility Study With Watchman Left Atrial Appendage Closure Technology). J Am Coll Cardiol. 2013 Jun 25;61(25):2551-6. doi: 10.1016/j.jacc.2013.03.035. Epub 2013 Apr 10. PMID 23583249
- [Background] Reddy VY, Holmes D, Doshi SK, Neuzil P, Kar S. Safety of percutaneous left atrial appendage closure: results from the Watchman Left Atrial Appendage System for Embolic Protection in Patients with AF (PROTECT AF) clinical trial and the Continued Access Registry. Circulation. 2011 Feb 1;123(4):417-24. doi: 10.1161/CIRCULATIONAHA.110.976449. Epub 2011 Jan 17. PMID 21242484
- [Background] Sick PB, Schuler G, Hauptmann KE, Grube E, Yakubov S, Turi ZG, Mishkel G, Almany S, Holmes DR. Initial worldwide experience with the WATCHMAN left atrial appendage system for stroke prevention in atrial fibrillation. J Am Coll Cardiol. 2007 Apr 3;49(13):1490-5. doi: 10.1016/j.jacc.2007.02.035. Epub 2007 Mar 21. PMID 17397680
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium (VARC)-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document (VARC-2). Eur J Cardiothorac Surg. 2012 Nov;42(5):S45-60. doi: 10.1093/ejcts/ezs533. Epub 2012 Oct 1. PMID 23026738
- [Background] Kefer J, Vermeersch P, Budts W, Depotter T, Aminian A, Benit E, Stammen F. Transcatheter left atrial appendage closure for stroke prevention in atrial fibrillation with Amplatzer cardiac plug: the Belgian Registry. Acta Cardiol. 2013 Dec;68(6):551-8. doi: 10.1080/ac.68.6.8000001. PMID 24579432
- [Background] Friberg L, Rosenqvist M, Lip GY. Evaluation of risk stratification schemes for ischaemic stroke and bleeding in 182 678 patients with atrial fibrillation: the Swedish Atrial Fibrillation cohort study. Eur Heart J. 2012 Jun;33(12):1500-10. doi: 10.1093/eurheartj/ehr488. Epub 2012 Jan 13. PMID 22246443
- [Derived] Teiger E, Eschalier R, Amabile N, Rioufol G, Ducrocq G, Garot P, Lepillier A, Bille J, Elbaz M, Defaye P, Audureau E, Le Corvoisier P; French Left Atrial Appendage Closure-2 registry (FLAAC-2) investigators. Left atrial appendage closure in very elderly patients in the French National Registry. Heart. 2024 Jan 29;110(4):245-253. doi: 10.1136/heartjnl-2023-322871. PMID 37813560